CLINICAL TRIAL: NCT07142629
Title: Selective Versus Non-selective Caries Excavation in MIH Affected Teeth: A Randomized Clinical Trial
Brief Title: Selective Versus Non-selective Caries Excavation in MIH Affected Teeth.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 413 - 2024; 20240457 . (Other Grant/Funding Number: Jordan University of Science and Technology)
Record Dates: First submitted 2025-05-07; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Molar Incisor Hypomineralisation; Dental Caries
Keywords: Molar Incisor Hypomineralisation; Selective caries removal; Non-selective caries removal
MeSH Terms: conditions — Molar Hypomineralization; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective caries removal (Experimental): Selective carious removal to firm dentine. Subsequently, 2 mm of Biodentine will be placed as a liner over the pulpal wall leaving the peripheries of the cavity available for bonding of the subsequent restoration.
  Interventions: Procedure: Selective caries removal
- Non-Selective caries removal (Experimental): Complete caries excavation will be done to hard scratchy dentine, with the aid of caries detector dye.If no pulp exposure is evident 2 mm of Biodentine will be placed and the cavity will be restored. If pulp exposure occurred, and it is bleeding normally and uniformly red with no zones of degeneration or necrosis then direct pulp capping will be attempted with Biodentine as a capping material. If no hemostasis is achieved, then the procedure will be modified to either partial pulpotomy, full pulpotomy or RCT depending on the clinical assessment.
  Interventions: Procedure: Non-Selective caries removal

INTERVENTIONS:
Procedure: Selective caries removal — Selective carious removal to firm dentine. Subsequently, 2 mm of Biodentine will be placed as a liner over the pulpal wall leaving the peripheries of the cavity available for bonding of the subsequent restoration.
  Arms: Selective caries removal
Procedure: Non-Selective caries removal — Complete caries excavation will be done to hard scratchy dentine, with the aid of caries detector dye.If no pulp exposure is evident 2 mm of Biodentine will be placed and the cavity will be restored. If pulp exposure occurred, and it is bleeding normally and uniformly red with no zones of degeneration or necrosis then direct pulp capping will be attempted with Biodentine as a capping material. If no hemostasis is achieved, then the procedure will be modified to either partial pulpotomy, full pulpotomy or RCT depending on the clinical assessment.
  Arms: Non-Selective caries removal

SUMMARY:
The aim of this study is to compare the clinical and radiographic outcomes of selective versus nonselective caries removal in MIH affected teeth with deep carious lesions using enhanced clinical protocols.

DETAILED DESCRIPTION:
The aim of this study is to compare the clinical and radiographic outcomes of selective versus nonselective caries removal in MIH affected teeth with deep carious lesions using enhanced clinical protocols.Cases will be collected from the undergraduate and postgraduate clinics over a 6 months' period according to predetermined inclusion criteria. Preoperative clinical and radiographic assessment will be conducted to MIH affected molars. MIH molars with deep caries (assymptomatic/ with symptoms of reversible pulpitis) will be randomly allocated for the choice of treatment with selective or non -selective caries excavation. Randomization of teeth between the 2 treatment groups will be performed using an online block randomization technique (block of 6) with the tooth as unit of randomization. Time taken for each procedure will be recorded by the research assistant each visit prospectively after achieving local anaesthesia till the end of procedure. Patients will be asked to rate their satisfaction with the received treatment on the end of treatment visit using a designed questionnaire. Clinical and radiographic success, and patient satisfaction will be evaluated at 6 and 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* The patient age <13 years old
* Non -contributory medical history
* Molar affected with MIH as per EAPD diagnostic criteria (White, creamy, or yellow to brownish opacities greater than one millimeter with/without postoperative enamel breakdown).
* Deep caries extending>= 2/3 of dentine but not exposing the pulp on the bitewing radiograph.
* The tooth should give positive response to cold sensibility testing.
* Clinical diagnosis of normal/ reversible pulpitis
* The tooth is restorable, probing pocket depth and mobility are within normal limits.
* No signs of pulpal necrosis including sinus tract or swelling
* No radiographic evidence of periapical changes indicative of apical periodontitis.

Exclusion Criteria:

* Medically compromised patient.
* Non-restorable tooth.
* Clinical diagnosis of irreversible pulpitis.
* Signs of pulpal necrosis including sinus tract or swelling.
* Teeth indicated for extraction for orthodontic reasons.
* Uncooperative children who could not be treated under local anesthesia.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Radiographic Success | 6,12 months
  No radiographic evidence of periapical changes indicative of apical periodontitis
Rate of Clinical Success | 6,12 months
  Absence of clinical symptoms of spontaneous pain, pain on percussion, pathologic mobility or abscess formation.,assessed through taking pain history and clinical examination.

SECONDARY OUTCOMES:
Patient acceptance of treatment | immediately following intervention, and at 6 and 12 months recall
  Self-reported child acceptance using questionnaire
Time taken for intervention | Perioperative/Periprocedural: from the time the child sits on the dental chair and until the intervention is completed.
  Time taken to perform intervention in minutes.
Child pain score | preoperatively and one week following the intervention
  Self-reported Child pain score preoperatively and one week after intervention, recorded on a scale of 0-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided